CLINICAL TRIAL: NCT04167319
Title: A Feasibility Study Investigating Chemotherapy-induced Neuropathy Using Multi-frequency Tactilometry and Patient-reported Outcomes (PRO)
Acronym: CINCAN-1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-088-2019
Record Dates: First submitted 2019-11-07; First posted 2019-11-18 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: CIPN; QST; Chemotherapy-induced Peripheral Neuropathy; Neurotoxic Chemotherapy; oxaliplatin; paclitaxel; Tactilometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected at baseline and after 3 courses of chemotherapy. Will be used for whole genome sequencing and specific findings will be correlated to CIPN QST Measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paclitaxel: Patients scheduled to receive paclitaxel as part of their standard treatment
  Interventions: Other: QST and PRO measurements during treatment
- Oxaliplatin: Patients scheduled to receive oxaliplatin as part of their standard treatment
  Interventions: Other: QST and PRO measurements during treatment

INTERVENTIONS:
Other: QST and PRO measurements during treatment — We will observe the natural course of CIPN using multiple measurements

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) is among the most feared side effects to cancer treatment. The development of CIPN can lead to discontinuation or omission of antineoplastic drugs, possibly affecting efficacy of cancer treatment. There is a lack of knowledge about the natural course of CIPN and to this date, there are no available methods for the early detection of CIPN. With no effective prevention or treatment options, the condition has severe impact on patient quality of life and healthcare expenditure.

This study will investigate the natural course of paclitaxel- and oxaliplatin induced peripheral neuropathy using novel diagnostic techniques. Multi-frequency vibrational technology has provided an objective method for the early detection of diabetic neuropathy. Our study will test the feasibility of this method within the field of clinical oncology and CIPN.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* A diagnosis of cancer.
* Fulfil the criteria for starting chemotherapy.
* Scheduled to undergo at least 4 courses of paclitaxel- or oxaliplatin-based chemotherapy.
* No prior paclitaxel, oxaliplatin or other neurotoxic chemotherapy.

Exclusion Criteria:

* Unable to complete PRO measures.
* Previous neurotoxic chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will invite patients to participate in conjuction with their standard treatment. Patients have been diagnosed with ovarian cancer or colorectal cancer and have been scheduled to adjuvant treatment or metastatic treatment with one of the applicable drugs.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Difference in VPT from baseline to 6 mo. | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in vibrograms from baseline compared to vibrograms after the end of the 6th course of chemotherapy or the last course of chemotherapy (if before course no. 6).
Difference in VPT from Baseline to 4 mo. | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in vibrograms from baseline compared to vibrograms after the end of the 4th course of chemotherapy or the last course of chemotherapy (if before course no. 4).

SECONDARY OUTCOMES:
Difference in PRO from baseline and during 1. course chemotherapy. | up to 5 days
  Difference in the NCCTG-CIPN Questionnaire from baseline compared to 4 days after initiation of chemotherapy course no. 1.
Difference in VPT from baseline and during 1. course chemotherapy | up to 5 days
  Difference in the Vibrograms from baseline compared to 4 days after initiation of chemotherapy course no. 1.
Difference in PRO from baseline to after chemotherapy course no. 3 | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in EORTC-QLQ-CIPN20 from baseline compared to after chemotherapy course no. 3.
Difference in PRO from baseline to after chemotherapy course no. 2 | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in EORTC-QLQ-CIPN20 from baseline compared to after chemotherapy course no. 2. Some patients receiving oxaliplatin will have 6 courses of planned chemotherapy or planned metastatic treatment, in this case comparison will be made after chemotherapy course no. 3.
Difference in VPT from baseline to af chemotherapy course no. 3 | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in the Vibrograms from baseline compared to after chemotherapy course no. 3.
Difference in VPT from baseline to af chemotherapy course no. 2 | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in the Vibrograms from baseline compared to after chemotherapy course no. 2. Some patients receiving oxaliplatin will have 6 courses of planned chemotherapy or planned metastatic treatment, in this case comparison will be made after chemotherapy course no. 3.
No. of discontinuations | through study completion, an average of 1 year and 6 months
  Number of patients not completing their planned courses of chemotherapy (reasons for discontinuation will be registered).
No. of dose reductions | through study completion, an average of 1 year and 6 months
  Number of patients that need reductions of chemotherapy dose (reasons will be registered)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology and Palliative Care, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No